CLINICAL TRIAL: NCT01981239
Title: Voice Analysis Using the LPC (Linear Predictive Coding)Method for the Prediction of Aspiration;Prospective, Positive-controlled, Single-blind, Single Cohort Clinical Study of Efficacy
Brief Title: Voice Analysis Using the LPC (Linear Predictive Coding)Method for the Prediction of Aspiration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participation over the long period
Sponsor: Ulsan University Hospital (Other)
Responsible Party: Principal Investigator, Chang Ho Hwang, Associate Professor, Ulsan University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: chhwang4
Record Dates: First submitted 2013-11-04; First posted 2013-11-11 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Deglutition Disorder
Keywords: voice analysis aspiration prediction
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LPC analysis group (Experimental): Voice sampling is executed before and immediately after drinking of 20ml N/S and linear voice analyses using LPC method are performed to calculate LPC index, residual variance, coefficiency mean, coeffiency variance, and coeffiency skewness.
  Interventions: Device: VFSS
- spectral analysis group (Active Comparator): Voice sampling is executed before and immediately after drinking of 20ml N/S and spectral voice analyses using Dr. Speech program are performed to calculate HNR (dB), RAP (%: Jitter), Mean and SD Fundamental Frequency (Hz: Fo), Shimmer (%) and SNR (dB).
  Interventions: Device: VFSS

INTERVENTIONS:
Device: VFSS — VFSS was perfomred one day before or after the voice sampling in the same patients according to the guideline of modified Longeman's protocol.

SUMMARY:
It was well known that aspiration is the primary cause of an aspiration pneumonia among the dysphagia patients.

In order to predict the degree of an aspitation,video-fluoroscopic-swallowing study and fiberoptic-endoscopic swallowing evaluation have been developed, but those evaluations are invasive and allowed only in a limited condition.

In this study, as a precedent study for the non-linear analysis, voice analysis using LPC method will be evaluated. The superiority of LPC method will be compared with a spectral analysis using Jitter and Simmer as a positive control.

This clinical study will be performed prospective, positive-controlled, single-blind (i.e. assessor-blind),and single cohort clinical trial for efficacy

ELIGIBILITY:
Inclusion Criteria:

* Patients who were referred for VFSS

Exclusion Criteria:

* Patients cannot phonate d/t tracheostomy
* Preexisting oro-laryngo-pharyngeal disease
* Patients cannot follow 1 step command
* Patients cannot maintain a phonation for 3 seconds
* Refusal of participation
* Patients who were not classified for the candidate by physicians
* Patients who coughs following drinking of 5ml normal saline

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
LPC index | one day before or after VFFS
  Voice sampling before and immediately after drinking of 20ml N/S and linear analysis using LPC method

SECONDARY OUTCOMES:
Spectral Analysis | one day before or after VFFS
  Voice sampling is performed before and immediately after drinking of 20ml N/S and HNR (dB), RAP (%: Jitter), Mean and SD Fundamental Frequency (Hz: Fo), Shimmer (%) and SNR (dB) are calculated using Dr. Speech program.
LPC anaysis | one day after or before VFSS
  Voice sampling is performed before and immediately after drinking of 20ml N/S and residual variance, coefficiency mean, coeffiency variance, and coeffiency skewness are computed using LPC analysis program.
Risk group | whithin one hour of VFSS
  According to Penetration-aspiration scale, patients are classified into high-risk patients (grade IV-VIII) and low-risk patients (grade I-III) by using the data derived from videofluoroscopic swallowing study

CONTACTS AND LOCATIONS:
Overall Officials: Chang Ho Hwang, M.D. & Ph.D., Study Director — Ulsan University Hospital; Hyungseob Han, M.Sc., Principal Investigator — University of Ulsan
Locations (1):
- Ulsan University Hospital, Ulsan, South Korea